CLINICAL TRIAL: NCT00547664
Title: Efficacy of Hylenex in the Treatment of Pain Among Hospice Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HPC Healthcare, Inc. (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HPC200710
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Pain Management
Keywords: Hylenex, time tagged pain pain reduction, hospice population
MeSH Terms: conditions — Agnosia | interventions — Morphine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: Hylenex recombinant , morphine, saline
- B (Placebo Comparator)
  Interventions: Drug: Hylenex recombinant , morphine, saline; Other: Saline

INTERVENTIONS:
Drug: Hylenex recombinant , morphine, saline — Subcutaneous infusion of morphine and hydromorphone (Dilaudid) with or without the preceded co-injection of Hylenex. Hospice patients include both home-bound patients as well as those under intensive care in hospice houses.
  Other Names: hyaluronidase human injection
Other: Saline — Subcutaneous infusion of morphine and hydromorphone (Dilaudid) with the preceded co-injection of saline.
  Other Names: Saline is used to determine the placebo effect.
  Arms: B

SUMMARY:
The overall aim of this study is to find out whether Hylenex recombinant (for short, Hylenex) in subcutaneous (SC) injection improves the speed and effectiveness of SC opioids in hospice patients. Specifically, this study proposes to compare the level of self-reported pain in hospice patients started on SC infusions of morphine and hydromorphone (Dilaudid) over the initial 8 hours of opioid infusion with and without the preceded co-injection of Hylenex. Hospice patients include both home-bound patients as well as those under intensive care in hospice houses.

DETAILED DESCRIPTION:
As of January 2009, 58 patients were recruited to the study as study subjects. Target goals for the study is to recruit 88 subjects with full and accurate information with about 44 patients in the Hylenex group and another group of subjects in the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant, non-lactating adults 18+ years enrolled in inpatient facilities at LifePath or Good Shepherd Hospice
2. Ability to provide informed consent; Patient has decision-making capacity (SPMSQ score 6+)
3. Ability to provide numerical report on pain level on pain scale
4. English-speaking
5. Pain not satisfactorily controlled with current meds -oral, topical, or rectal; Pain level greater than 3 at admission on a 0-10 scale
6. Able to self-administer bolus dose or ask someone to hit bolus button
7. Estimated life expectancy of 3 days or more
8. Patients appropriate for continuous SC infusion with either morphine or hydromorphone.

Exclusion Criteria:

1. History of allergy or hypersensitivity to Hylenex or any components of product
2. Patients on infusion therapy for pain management up to 14 days prior to entering inpatient facilities.
3. Patients who are actively dying identified by any of the following physical signs and symptoms:

   1. non-communicative or unresponsiveness; b) confusion/disorientation about time, place, and people; c) significant chest congestion with gurgling sounds; d) restless and repetitive motions; e) little or no food or fluid intake; f) minimal urine output and g) different breathing pattern, i.e., shallow rapid breaths with period of no breathing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the sum of 7 pain intensity differences (SPID) computed from 8 observations of pain during the 8-hour period. | For a period of 8 hours from start to finish

SECONDARY OUTCOMES:
The secondary outcome measure will be the sum of distress level differences (SDLD), sum of relief level differences (SRLD), and sum of bolus attempts (SBAM) made during the same 8-hour period. | For a period of 8 hours from start to finish
The mean number of bolus attempts made over the 8-hour period between experimental and control groups. | The bolus attempts will be observed for the 8-hour period from start to finish.

CONTACTS AND LOCATIONS:
Overall Officials: Sehwan Kim, Ph.D, Study Director — HPC Healthcare, Inc.
Locations (3):
- United States (3):
  - Good Shepherd Hospice, Lakeland, Florida
  - LifePath Hospice, Inc., Tampa, Florida
  - HPC Healthcare, Inc., Temple Terrace, Florida